CLINICAL TRIAL: NCT04010422
Title: Evaluating the Ocular Function of Adults With Autism Spectrum Disorder: Interrelationship Between Blinking Reflex and Cornea Innervation.
Brief Title: Ocular Function in Autism Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904121RINC
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Autism; Ocular Surface Disease
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD group: Inclusion Criteria:
  1. Having a clinical diagnosis of autism spectrum disorder
  2. Aged over 20 years; able to read and sign an informed consent form.
  3. Clear conscious and can follow the instruction of opening eyes and movement toward all direction.
  Exclusion Criteria:
  1. Unable to cooperate with the examinations.
  2. Younger than 20 years old
  Interventions: Diagnostic Test: no intervention
- TD Group: Inclusion Criteria:
  1. Aged over 20 years; able to read and sign an informed consent form.
  2. Clear conscious and can follow the instruction of opening eyes and movement toward all direction.
  Exclusion Criteria:
  1. Unable to cooperate with the examinations.
  2. Younger than 20 years old.
  3. Having a clinical diagnosis of autism spectrum disorder
  Interventions: Diagnostic Test: no intervention

INTERVENTIONS:
Diagnostic Test: no intervention — no intervention

SUMMARY:
This study will investigate the visual function in individuals with ASD, with a particular focus on the ocular surface condition and visual function assessment.

DETAILED DESCRIPTION:
Anomalies in visual information processing can have a major effect on the life quality of individuals with autism spectrum disorders (ASD), including eye gaze abnormality, higher frequency of refractive errors (e.g., astigmatism, hypermetropia, and anisometropia), strabismus, abnormal blinking rate, disturbed eye movements that may be associated with or aggravated social communication deficits of ASD. However, little is known about the ocular surface conditions. This study will investigate the visual function in individuals with ASD, with a particular focus on the ocular surface condition. We plan to recruit 50 adults with ASD and 50 age-/sex-matched typically developing controls in this project, and perform visual function assessment.

ELIGIBILITY:
ASD group:

Inclusion Criteria:

1. Having a clinical diagnosis of autism spectrum disorder
2. Aged over 20 years; able to read and sign an informed consent form.
3. Clear conscious and can follow the instruction of opening eyes and movement toward all direction.

Exclusion Criteria:

1. Unable to cooperate with the examinations.
2. Younger than 20 years old.

TD group:

Inclusion Criteria:

1. Aged over 20 years; able to read and sign an informed consent form.
2. Clear conscious and can follow the instruction of opening eyes and movement toward all direction.

Exclusion Criteria:

1. Unable to cooperate with the examinations.
2. Younger than 20 years old.
3. Having a clinical diagnosis of autism spectrum disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an observation study. We will recruit 50 adults with autism spectrum disorder aging over 20 years old from the Psychiatry Department, National Taiwan University Hospital. We will also recruit 50 adults without autism spectrum disorder aging over 20 years old from the Ophthalmology Department, National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
cornea innervation | 30 min
  The participants will undergo HRT in vivo confocal microscopy. It is a laser scanning confocal microscope, operating by scanning a 670 nm laser beam in a raster pattern over the field of view. The system uses a high numerical aperture 63x objective lens (0.9 NA), and produces images with high contrast and better axial resolution (7.6 µm) than other in vivo confocal systems (9 µm for the TSCM and 24 µm for the Confoscan). The HRT-RCM provides new built-in software for 3D imaging of the corneal structure. Quantitative imaging of the subbasal nerve plexus could be per-formed by CCMetrics system, a custom software program developed at the University of Manchester.
Blinking reflex | 30 min
  Blinking rates manually calculated by two different research personnel and Tobii Pro X3-120 under two conditions: viewing preset film on the laptop and casual conversation with interviewer.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ling Chien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu CS, Tsai HJ, Chien YL, Gau SS. All-Cause Mortality and Specific Causes of Death in Autism: A Nationwide Analysis. Autism Adulthood. 2025 Feb 5;7(1):81-92. doi: 10.1089/aut.2023.0103. eCollection 2025 Feb. PMID 40151655